CLINICAL TRIAL: NCT05965986
Title: Preoperative Patient Education and Rehabilitation Program for a Total Shoulder Arthroplasty Surgery: a Pilot Randomized Control Trial
Brief Title: Preoperative Rehabilitation and Education Program
Acronym: PREPS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Western University, Canada (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Joy MacDermid, Professor, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 120163
Record Dates: First submitted 2023-07-07; First posted 2023-07-28 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Shoulder Arthritis; Patient Education; Prehabilitation; Shoulder Arthroplasty
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard of Care Group (No Intervention): A group consisting of the current standard of care at HULC, which is a WebEx pre-operative education class lead by a physiotherapist and occupational therapist.
- Online only (Experimental): a group consisting of an online pre-rehabilitation program 6 weeks before surgery
  Interventions: Other: Experimental: PREPS only
- Online and PT (Experimental): a group consisting of an online pre-rehabilitation program 6 weeks before surgery + therapist
  Interventions: Other: Experimental: PREPS and therapy

INTERVENTIONS:
Other: Experimental: PREPS only — Participants will be guided through an education program and exercise program that will cover topics. Participants will have flexibility as to when and how often then need to review material. Participants will be directed to completed on-screen interactive quizzes to re-enforce learning. Participants are encouraged to pose any questions regarding the material they are learning within the education modules to the research team for further clarification.
  The intervention group will be asked to participate in the program (6 weeks), but after their surgery, they will not be asked to continue the education or exercise program. However, they will be tracking their activity and adherence to physical therapy through a log for one year post-operative.
  Arms: Online only
Other: Experimental: PREPS and therapy — Participants will be guided through an education program and exercise program that will cover topics. Participants will have flexibility as to when and how often then need to review material. Participants will be directed to completed on-screen interactive quizzes to re-enforce learning. Participants are encouraged to pose any questions regarding the material they are learning within the education modules to the research team for further clarification.
  The intervention group will be asked to participate in the program (6 weeks), but after their surgery, they will not be asked to continue the education or exercise program. However, they will be tracking their activity and adherence to physical therapy through a log for one year post-operative. In addition, participants will have a therapist call on week 2 and 4 of the program and then one week after surgery to check in and ensure the patient is meeting all milestones and answer any questions.
  Arms: Online and PT

SUMMARY:
Shoulder problems affect many Canadians yearly. While surgery is one of the best treatments for shoulder problems, patients are unaware about shoulder replacement surgeries, the exercises needed after surgery and how to safely recover from the surgery without having another injury. Uncertainties about the surgery and recovery process can further cause post-surgery problems such as: pain, anxiety and re-injury. While some healthcare centers offer an in- class program to educate patients before surgery, some patients face issues with distance or transportation, and cannot regularly meet their doctor to address all their concerns. This project aims to create an online educational program that will teach patients through online videos and educational materials before they go into shoulder replacement surgery. By creating online modules, it can increase the accessibility for home use, and prepare patients on topics such as: their concerns about the surgery and proper exercises they can expect after surgery for a safe recovery. The aim is to study three groups of patients before surgery; 1. a group consisting of an online pre-rehabilitation program 6 weeks before surgery, 2. a group consisting of an online pre-rehabilitation program 6 weeks before surgery + therapist or 3. A group consisting of the current standard of care, which is a WebEx pre-operative education class lead by a physiotherapist and occupational therapist. Researchers will monitor all groups on their recovery before and after surgery. This will provide another alternative to informing patients before surgery and help them to prepare better for surgery. The online modules will contribute to improving the care in Southern Ontario and eventually be used for future care across Canada.

DETAILED DESCRIPTION:
A total shoulder replacement is a common procedure to help those with shoulder osteoarthritis improve their quality of life. There is a lack of quality research on the effectiveness of prehabilitation and education on pain, function, and quality of life in patients undergoing this procedure. Researchers have developed a comprehensive, patient-centered program that combines exercise, preparedness for surgery, motivational interviewing, and pain management principles, in collaboration with patient partners on the wait list for a shoulder replacement, transdisciplinary healthcare team (i.e., surgeons, physiotherapists, occupational therapists, and rehabilitation researchers), and current scientific literature. This patient-centered program has the potential to improve postoperative pain, function, and patient-oriented outcomes, decrease postoperative opioid use and short and long-term healthcare costs. This pilot randomized controlled trial will evaluate feasibility and satisfaction of the program for individuals undergoing a shoulder replacement. Participants (n=90) undergoing a shoulder replacement will be randomized into 1) 6-week online pre-rehab and education program, 2) 6-week online pre-rehab and education program with a therapist or 3) standard of care group. The intervention groups will be delivered virtually with an online program of modules and a written handbook for participants. Participants in the standard of care group will receive usual care. Outcomes will be assessed at baseline and 1 day before surgery, then post-operatively at 6 weeks, 3 months, 6 months and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Over the age of 18 years old
* Patients who have consented for a total shoulder arthroplasty or reverse shoulder arthroplasty surgery at HULC.
* Date of surgery must be no shorter than 9 weeks, to ensure time for baseline measures
* Speaks and reads in English unless can provide a translator
* Able to provide informed consent.
* Willing to participate in study procedures for at least 1 year post-surgery.

Exclusion Criteria:

* Patients who have consented for a hemi-arthroplasty surgery
* Patients who have been consented less than 8 weeks before surgery
* Any contraindications to exercise

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Recruitment Rate log | 6 months
  We will proceed with the larger trial if we are able to recruit 90 participants within 6 months, and if 50% of eligible participants consent to participate.
Adherence Rate log | 6 months
  Adherence to the education program will be considered adequate if 80% of all participants in the intervention groups complete the full online program and report it on the log. Exercise programs will be considered adequate if 60% of participants in the intervention groups report exercise at least 3 times per week.
Content Acceptability - visual analog scale | 12 months
  Content acceptability will be assessed using a visual analog scale (VAS), where acceptability will be considered adequate if 60% of participants found the treatment useful and helpful with a score of 7/10.
Study Acceptability - visual analog scale | 12 months
  Similarly, if 60% of participants found the treatment delivery acceptable, and reported being likely to use this treatment again and recommend it to others with a VAS score of 7/10, the format will be considered acceptable.
Treatment Fidelity checklist | 12 months
  if 80% of phone calls were documented accurately and able to meet the criteria of the checklist by the therapist, fidelity will be considered acceptable.

SECONDARY OUTCOMES:
5-level EQ-5D version | 12 months
  General Health Status
Simple Shoulder Test | 12 months
  functional outcome measure
Single Assessment Numeric Evaluation | 12 months
  functional outcome measure
Range of motion | 12 months
  shoulder movement
Surgical Satisfaction Questionnaire | 3 months
  satisfaction with surgery
Decisional Regret | 3 months
  decisional conflict with surgery or the preparation
Adherence to rehabilitation | 12 months
  adherence to a post-surgery rehabilitation program
PASS | 12 months
  Single item to understand people's satisfaction with their current health condition
Shoulder Pain and Disability Index | 12 months
  shoulder pain and function for shoulder conditions

CONTACTS AND LOCATIONS:
Overall Officials: Joy MacDermid, PhD, Principal Investigator — Western University, Canada
Locations (1):
- Roth | McFarlane Hand and Upper Limb Center, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Furtado R, MacDermid JC, Bryant D, Faber KJ. Preoperative rehabilitation and education program for surgery (PREPS): A pilot randomized control trial protocol. Hand Ther. 2025 Jun 20;30(4):200-207. doi: 10.1177/17589983251345393. eCollection 2025 Dec. PMID 40547196